CLINICAL TRIAL: NCT03265821
Title: Influence of Smoking on Periodontal Healing One Year After Active Treatment
Status: Completed | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Kristina Edman, Reg dental hygienist, medical doctor, Dalarna County Council, Sweden
Other Study IDs: Smoking periodontal healing
Record Dates: First submitted 2017-08-28; First posted 2017-08-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Periodontal Diseases; Smoking
Keywords: Smoking; Periodontal treatment; Periodontal disease; Healing
MeSH Terms: conditions — Periodontal Diseases; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Healing after treatment

SUMMARY:
The aim of this study was to investigate whether cigarette smoking had any impact on the clinical outcomes 1 year after active periodontal treatment. Eligible for the study were 5680 individuals 20-85 years, referred to the specialised clinic for periodontal treatment at Gävle County Hospital between the years of 1980 and 2015. Before examination, all individuals filled in a questionnaire regarding their medical health, medication and smoking habits.

Excluded were edentulous individuals and where clinical data 1-year after active treatment, or smoking habits were missing (n=1453). Complete data for analyses was available for 4227 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals referred to a specialist clinic for periodontal treatment

Exclusion Criteria:

* edentulous individuals

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals 20-85 years, referred to the specialised clinic for periodontal treatment at Gavle County Hospital, Sweden between the years of 1980 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 4227 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | 1 year
  Probing pocket depth